CLINICAL TRIAL: NCT04421729
Title: SoCal Savvy: Testing Savvy Caregiver in a Racially and Ethnically Diverse Sample in
Brief Title: SoCal Savvy: Testing Savvy Caregiver in a Racially and Ethnically Diverse Sample in Southern California
Acronym: SoCalSavvy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Maria P. Aranda, Associate Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 5356000538
Record Dates: First submitted 2020-06-02; First posted 2020-06-09 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Caregiver Burnout; Psychological Distress
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will not have previous knowledge of the respondent's interventional group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Savvy Caregiver Program (Active Comparator): Savvy Caregiver Program, 6 weekly sessions, group treatment, addressing educational, informational, and psychosocial issues and community resources.
  Interventions: Behavioral: Group sessions over 6 weeks
- Savvy Express (Active Comparator): Savvy Express, 3 weekly sessions, group treatment, addressing educational, informational, and psychosocial issues and community resources.
  Interventions: Behavioral: Group sessions over 3 weeks

INTERVENTIONS:
Behavioral: Group sessions over 3 weeks — Informational and educational group-mediated program for family members caring for a person living with dementia; 6 sessions.
  Arms: Savvy Express
Behavioral: Group sessions over 6 weeks — Informational and educational group-mediated program for family members caring for a person living with dementia; 3 sessions.
  Arms: Savvy Caregiver Program

SUMMARY:
The investigators will conduct a hybrid efficacy-effectiveness trial intended to address these gaps by testing the efficacy-effectiveness of two multi-family group interventions, and on 250 English-speaking adults: Savvy Caregiver Express™ (3-session, newly piloted in Los Angeles County for feasibility) and Savvy Caregiver Program (original 6-session evidenced-based intervention), across post-intervention, 3- and 6-months.

DETAILED DESCRIPTION:
A number of epidemiological studies, systematic reviews, and consensus reports highlight the importance of non-pharmacological, sociobehavioural interventions to address the health, psychological, and social effects of caregiving for persons living with dementia, and the need for tangible information and resources.

The investigators will conduct a hybrid efficacy-effectiveness trial intended to address these gaps by testing the efficacy-effectiveness of two multi-family group interventions, and on 250 English-speaking adults: Savvy Caregiver Express™ (3-session, newly piloted in Los Angeles County for feasibility) and Savvy Caregiver Program (original 6-session evidenced-based intervention), across post-intervention, 3- and 6-months. It is hypothesized that no differences (comparable effects) between the programs in their efficacy/effectiveness and moderating conditions.

Focus groups (~25 participants) will be conducted to ascertain program acceptability and satisfaction.

The analyses will include a multiple linear mixed-effects modeling for our trial outcomes, and thematic analyses for our focus group interview data.

ELIGIBILITY:
Inclusion Criteria:

* English- speaking women and men age 18 or older who care for or provide assistance to someone with dementia

Exclusion Criteria:

* Caregivers who have sensory or physical conditions that interfere with participation in an on-site, group-administered activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | up to 7 months
  caregiver depressive symptoms
Generalized Anxiety Disorder (GAD-7) | up to 7 months
  caregiver anxiety symptoms
Revised Memory and Behavior Problems Checklist (RMBPC) | up to 7 months
  caregiver reactivity to family member's memory/behavior problems

SECONDARY OUTCOMES:
Caregiver Competence Scales | up to 7 months
  measures caregiver skills, mastery, competence, management of the situation based on the Caregiver Competence, Management and Meaning Scales
Medical Outcomes Study Social Support Survey (MOS) | up to 7 months
  Measures caregiver social support using the MOS scale
Intent to Institutionalize | up to 7 months
  TA one-item measure that assesses if the caregiver intends to institutionalize the family member in the next 6 months
Family Members Activities of Daily Living (ADL) | up to 7 months
  measures family member's activities of daily living using the Katz ADL scale
Family Members Instrumental Activities of Daily Living (IADL) | up to 7 months
  measures family member's activities of daily living using the Lawton IDL scale

OTHER OUTCOMES:
Caregiver Satisfaction | up to 7 months
  This is a measure developed for this specific study to ascertain the study participant's satisfaction with the intervention itself.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No